CLINICAL TRIAL: NCT01252121
Title: Residence Time Evaluation of Systane Ultra Lubricant Eye Drops vs. Hialid and Saline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RDG-10-275; CS-10-01 (Other: Xiamen University)
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-05

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye; Ocular Retention Time
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Systane, Hialid, Unisol (Other): 1 drop Systane in study eye at Visit 2, 1 drop Hialid in study eye at Visit 3, 1 drop Unisol in study eye at Visit 4, with a minimum of 24 hours between each visit.
  Interventions: Other: Systane Ultra Lubricant Eye Drops; Other: Hialid 0.1 Artificial Tears Eye Drops; Other: Unisol 4 Saline Solution
- Systane, Unisol, Hialid (Other): 1 drop Systane in study eye at Visit 2, 1 drop Unisol in study eye at Visit 3, 1 drop Hialid in study eye at Visit 4, with a minimum of 24 hours between each visit.
  Interventions: Other: Systane Ultra Lubricant Eye Drops; Other: Hialid 0.1 Artificial Tears Eye Drops; Other: Unisol 4 Saline Solution
- Hialid, Systane, Unisol (Other): 1 drop Hialid in study eye at Visit 2, 1 drop Systane in study eye at Visit 3, 1 drop Unisol in study eye at Visit 4, with a minimum of 24 hours between each visit.
  Interventions: Other: Systane Ultra Lubricant Eye Drops; Other: Hialid 0.1 Artificial Tears Eye Drops; Other: Unisol 4 Saline Solution
- Hialid, Unisol, Systane (Other): 1 drop Hialid in study eye at Visit 2, 1 drop Unisol in study eye at Visit 3, 1 drop Systane in study eye at Visit 4, with a minimum of 24 hours between each visit.
  Interventions: Other: Systane Ultra Lubricant Eye Drops; Other: Hialid 0.1 Artificial Tears Eye Drops; Other: Unisol 4 Saline Solution
- Unisol, Systane, Hialid (Other): 1 drop Unisol in study eye at Visit 2, 1 drop Systane in study eye at Visit 3, 1 drop Hialid in study eye at Visit 4, with a minimum of 24 hours between each visit.
  Interventions: Other: Systane Ultra Lubricant Eye Drops; Other: Hialid 0.1 Artificial Tears Eye Drops; Other: Unisol 4 Saline Solution
- Unisol, Hialid, Systane (Other): 1 drop Unisol in study eye at Visit 2, 1 drop Hialid in study eye at Visit 3, 1 drop Systane in study eye at Visit 4, with a minimum of 24 hours between each visit.
  Interventions: Other: Systane Ultra Lubricant Eye Drops; Other: Hialid 0.1 Artificial Tears Eye Drops; Other: Unisol 4 Saline Solution

INTERVENTIONS:
Other: Systane Ultra Lubricant Eye Drops — One drop in study eye, one time, during office visit.
Other: Hialid 0.1 Artificial Tears Eye Drops — One drop in study eye, one time, during office visit.
Other: Unisol 4 Saline Solution — One drop in study eye, one time, during office visit.

SUMMARY:
The purpose of this study is to evaluate the ocular retention time of Systane Ultra compared to Hialid and saline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mild to moderate dry eye as defined in the protocol.
* Able and willing to follow instructions.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any medical condition that may affect the results of the study.
* History or evidence of ocular or intraocular surgery within the past six months.
* History of intolerance or hypersensitivity to any component of the study medications.
* Use of concomitant topical ocular medications during the study period.
* Ocular conditions that may preclude safe administration of the test article.
* Unwilling to discontinue contact lens wear during the study period.
* Participation in an investigational drug or device study within 30 days of enrollment.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Ocular surface residence time | Time to event
  Ocular surface residence time is defined as the time for fluorescence intensity to return to baseline value after a drop of ophthalmic dye is instilled in the study eye. Dye retention will be measured with a fluorophotometer.